CLINICAL TRIAL: NCT05110976
Title: Phase I, Randomised, Blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD8630 in Healthy Adult Subjects (Part A) and Adults With Asthma on Medium to High Dose Inhaled Corticosteroids and Long-acting Beta-agonists (Part B)
Brief Title: A Study to Investigate the Safety, Tolerability and Effects of AZD8630 in Healthy Subjects and Subjects With Asthma on Inhaled Corticosteroids and Long-acting Beta-agonists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: D6830C00001; 2021-004000-18 (EudraCT Number)
Record Dates: First submitted 2021-10-28; First posted 2021-11-08 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Asthma
Keywords: Healthy adult participants; Healthy participants of Chinese and Japanese ethnicity; Corticosteroids Beta-agonists; Multiple ascending dose; Single ascending dose
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A of the study is single-blind, and Part B of the study is double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part A1: SAD (AZD8630) (Experimental): Healthy participants will receive single inhaled doses 1 to 5 of AZD8630.
  Interventions: Drug: AZD8630
- Part A1: IV (AZD8630) (Experimental): Healthy participants will receive a single IV dose of AZD8630.
  Interventions: Drug: AZD8630
- Part A1: IV (Placebo) (Placebo Comparator): Healthy participants will receive single IV dose of Placebo.
  Interventions: Drug: Placebo
- Part A2: SAD (AZD8630) (Experimental): Healthy participants of Chinese and Japanese ethnicity will receive single inhaled dose 5 of AZD8630.
  Interventions: Drug: AZD8630
- Part A3: MAD (AZD8630) (Experimental): Healthy participants will receive once daily inhaled doses 3, 4, and 5 of AZD8630.
  Interventions: Drug: AZD8630
- Part A4: MAD (AZD8630) (Experimental): Healthy participants of Chinese and Japanese ethnicity will receive once daily inhaled dose 5 of AZD8630.
  Interventions: Drug: AZD8630
- Part A: SAD (Placebo) (Placebo Comparator): Healthy participants and healthy participants of Chinese and Japanese ethnicity will receive single inhaled doses of placebo.
  Interventions: Drug: Placebo
- Part A: MAD (Placebo) (Placebo Comparator): Healthy participants and healthy participants of Chinese and Japanese ethnicity will receive once daily inhaled dose of placebo.
  Interventions: Drug: Placebo
- Part B (AZD8630) (Experimental): Participants with asthma will be randomized to one of 3 inhaled dose levels 3, 6, and 7 of AZD8630 once daily.
  Interventions: Drug: AZD8630
- Part B (Placebo) (Placebo Comparator): Participants with asthma will receive once daily inhaled dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8630 — Participants will receive Inhaled or IV doses of AZD8630 as per the arm they are assigned.
  Arms: Part A1: IV (AZD8630); Part A1: SAD (AZD8630); Part A2: SAD (AZD8630); Part A3: MAD (AZD8630); Part A4: MAD (AZD8630); Part B (AZD8630)
Drug: Placebo — Participants will receive Inhaled or IV doses of placebo as per the arm they are assigned.
  Arms: Part A1: IV (Placebo); Part A: MAD (Placebo); Part A: SAD (Placebo); Part B (Placebo)

SUMMARY:
This is a first in human (FIH) clinical study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD8630 in healthy adults (Part A) and adult asthma patients on medium to high dose inhaled corticosteroids / Long-acting beta-agonists (Part B)

DETAILED DESCRIPTION:
The study is divided in 2 parts, A and B.

Part A will be conducted in healthy adults, whereas Part B will be conducted in adult asthma patients on medium/high dose inhaled corticosteroids (ICS)/long-acting beta-agonists (LABA) to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of AZD8630 by dry powder inhaler (DPI) administration. Part A includes the assessment of the PK and safety of intravenous (IV) AZD8630. Part A consists of single ascending dose (SAD) and multiple ascending dose (MAD) cohorts in sequential order and Part B will be evaluating multiple dose levels.

Part A: This part will consist 4 sub-parts and will include healthy participants and healthy participants of Chinese and Japanese ethnicity. These participants will randomized to receive AZD8630 and to receive placebo.

* Sub-Part A1, SAD in healthy participants (one cohort in Sub-Part A1 will receive IV AZD8630 [IV formulation])
* Sub-Part A2, SAD in healthy participants of Chinese and Japanese ethnicity
* Sub-Part A3, MAD in healthy participants
* Sub-Part A4, MAD in healthy participants of Chinese and Japanese ethnicity

Part B: Adult asthma patients will be randomized to one of 3 inhaled dose levels of AZD8630 or placebo.

The expected duration of study participation for each participants in the part A is up to 87 days, and each patients in the Part B is up to 70 days.

ELIGIBILITY:
Inclusion Criteria:

Part A (Healthy participants):

1. Healthy participants aged 18 to 55 years, inclusive:

   1. Japanese participants must be aged 20 to 55 years, inclusive
   2. Chinese participants must be aged 18 to 45 years, inclusive
2. Females must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test on admission to the Clinical Unit, must not be lactating, and must be of non childbearing potential, confirmed at the Screening Visit
3. Have a body mass index (BMI) between 18 and 30 kg/m^2 inclusive and weigh at least 45 kg.
4. Healthy participant must have a forced expiratory volume in 1 second (FEV1) ≥ 80% of the predicted value regarding age, height, gender, and ethnicity at the Screening Visit.
5. Male participants and their women of childbearing potential partners (WOCPB) should be willing to use highly effective contraception measures and male participants should refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the study Follow up Visit.
6. Part A2 and Part A4 (Chinese population only): Chinese participants must have been born in China, have all parents and grandparents of Chinese origin, and not have lived outside of China for more than 10 years.
7. Part A2 and Part A4 (Japanese population only): Japanese participants must have been born in Japan, have all parents and grandparents of Japanese origin, and not have lived outside of Japan for more than 10 years.

Part B (Participants with Asthma):

1. Male and female including WOCBP participants with asthma aged 18 to 75 years inclusive, with suitable veins for cannulation or repeated venipuncture.
2. Have a BMI between 18 and 35 kg/m^2 inclusive and weigh at least 45 kg.
3. Confirmed physician-led diagnosis of asthma for > 6 months before the Screening Visit.
4. Any of the following assessments within the last 10 years to confirm variable airflow obstruction: Variability between clinic visits: FEV1 > 12% and 200 mL; Response to 4 weeks' anti-inflammatory therapy: FEV1 > 12% and 200 mL; Exercise challenge test: FEV1 fall > 10% and 200mL; Methacholine challenge test: FEV1 ≥ 20% fall at < 8 mg/mL; Indirect challenge test: FEV1 ≥ 15% fall; Or in the screening period: Variability between clinic visits: FEV1 > 12% and 200 mL; Peak expiratory flow rate (PEFR) for 2 weeks during run-in: PEFR average daily variability > 10%.
5. Pre-bronchodilator FEV1 ≥ 40% and < 85% predicted at the Screening Visit.
6. Have a fractional exhaled nitric oxide (FeNO) of ≥ 35 ppb at the Screening Visit and ≥ 30 ppb at randomisation.
7. Asthma Control Questionnaire -5 score of ≥ 0.75 and ≤ 3.0 at screening.
8. During 7 consecutive days within screening, immediately prior to randomisation demonstrates ≥ 65% adherence to each of the following:

   1. Once daily home FeNO
   2. Twice daily home spirometry measurements
   3. Twice daily entries in the eDiary
9. Females must have a negative serum pregnancy test at the Screening Visit. Additionally, WOCBP must have a negative urine pregnancy test at Visit 2 (prior to randomisation) and must not be lactating.
10. Male participants and their WOCBP partners should be willing to use highly effective contraception measures and male participants should refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the study Follow-up Visit.
11. WOCBP must be willing to use highly effective contraception measures from the first day of dosing until 3 months after the study Follow up Visit.

Exclusion Criteria:

Part A (Healthy participants)

1. History of following: any clinically important disease or disorder; any upper or lower respiratory tract infection during screening period; active tuberculosis or current positive result for Interferon gamma release assay at screening; clinically significant history of atopy or allergy to common allergens including house dust mite and pollens, or a history of childhood asthma.
2. Active or previous hepatitis B, hepatitis C, or Human immunodeficiency virus at the Screening Visit, and other latent or chronic infections.
3. History of severe COVID-19 (Coronavirus disease 2019) infection requiring hospitalization
4. SARS-CoV-2 (Severe acute respiratory syndrome coronavirus 2) first vaccination within 30 days prior to screening.
5. SARS-CoV-2 second or booster vaccination within 10 days of screening.
6. Unwilling to defer SARS-CoV-2 vaccination during the study period.
7. History of cancer within last 10 years (20 years for breast cancer) except for basal and squamous cell carcinoma of skin or in situ carcinoma of cervix treated and considered cured. Any history of lymphoma is not allowed.
8. Have received live or live attenuated vaccine in 4 weeks prior to randomisation.
9. History of acquired or inherited immunodeficiency disorders including but not limited to HIV, COVID-19, or taking immune replacement therapy.
10. C-reactive protein above upper limit of laboratory reference range
11. Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results and abnormal vital signs at the Screening Visit.
12. Current smokers or those who have smoked or used nicotine or inhalational cannabis/marijuana products. History of alcohol abuse or drug abuse.
13. Use of any prescribed or nonprescribed medication during the 2 weeks prior to the first administration of investigational medicinal product.
14. Has received another new chemical entity.
15. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8630.
16. History of anaphylaxis to any previous biological therapy.
17. Participants who have previously received AZD8630.

Part B (Participants with Asthma):

1. History of following: any clinically important disease or disorder; any chronic respiratory disorders (except asthma) such as Chronic obstructive pulmonary disease, bronchiectasis, or IPF; clinically significant lower respiratory tract infection not resolved within 4 weeks prior to screening.
2. Acute exacerbation of asthma requiring hospitalisation and/or attendance at an emergency department and/or systemic corticosteroids within 6 weeks of randomisation.
3. History of active TB or a current positive result for IGRA at screening.
4. History of severe COVID-19 infection requiring hospitalisation.
5. SARS-CoV-2 first vaccination within 30 days prior to screening.
6. SARS-CoV-2 second or booster vaccination within 10 days of screening.
7. Confirmed COVID-19 infection during screening, prior to randomisation.
8. History of cancer within the last 10 years (20 years for breast cancer) except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured. Any history of lymphoma is not allowed.
9. Have received live or live attenuated vaccine in the 4 weeks prior to randomisation.
10. C-reactive protein above the upper limit of laboratory reference range at screening.
11. Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results, and abnormal vital signs at the Screening Visit.
12. Current smokers or those who have smoked or used nicotine or inhalational cannabis/marijuana products. History of alcohol or drug abuse.
13. Positive screen for drugs of abuse or cotinine (nicotine) prior to randomisation.
14. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks before first administration of study drug.
15. Use of any prescribed or nonprescribed medication during the 2 weeks prior to the first administration of study drug.
16. Use of following medicines within specified time before Screening: (a) Any biologics for asthma within 6 months prior to Screening; (b) Systemic or intranasal steroids within 4 weeks prior to Screening; (c) Xanthines, anticholinergics, or cromoglycate within 1 week prior to Screening; (d) Short acting bronchodilator other than for rescue and within 12 hours prior to Screening and Day -1 assessments.
17. History of anaphylaxis or ongoing clinically important serious allergy, or history of hypersensitivity or anaphylaxis to drugs with a similar chemical structure or class to AZD8630.
18. History of anaphylaxis to any previous biological therapy.
19. Pregnancy or intention to become pregnant during course of study, breastfeeding, or unwillingness to use a highly effective method of contraception throughout study in female participants of childbearing potential or lactating woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Number of participants with adverse events | Until Follow-up (FU) Visit/Early Termination (ET) Visit (Part A: 7-day post-dose for SAD; 10-day post-last dose for MAD) and Part B: Until FU Visit/ET Visit (10-day post-last dose)
  Safety and tolerability of inhaled AZD8630 in healthy participants and participants with asthma will be assessed.
Part A (IV cohort): Time to reach maximum observed concentration (tmax) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  tmax of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed
Part A (IV cohort): Time of last observed quantifiable concentration (tlast) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  tlast of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed
Part A (IV cohort): Maximum observed serum (peak) drug concentration (Cmax) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  Cmax of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Partial area under the serum concentration-time curve from 0 to time 24 hours post-dose [AUC(0-24)] of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  AUC(0-24) of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Area under the serum concentration curve from zero to the last quantifiable concentration (AUClast) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  AUClast of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Area under serum concentration-time curve from zero to infinity (AUCinf) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  AUCinf of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Terminal rate constant (λz) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  λz of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  t1/2λz) of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Mean residence time of the unchanged drug in the systemic circulation (MRTinf) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  MRTinf of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Total body clearance of drug from serum after IV administration (CL) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  CL of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV cohort): Volume of distribution at steady state (Vss) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  Vss of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV Cohort): Volume of distribution of drug from serum after IV administration (Vz) of AZD8630 | Pre-dose and Post-dose on Days 1 to 4 and Follow-up Visit/ET Visit (7-day post-dose)
  Vz of AZD8630 following IV administration of single dose of AZ8630 in healthy participants will be assessed.
Part A (IV Cohort): Number of participants with adverse events | Until Follow-up (FU) Visit/Early Termination (ET) Visit (7-day post-dose)
  Safety and tolerability of IV AZD8630 in healthy participants will be assessed.

SECONDARY OUTCOMES:
Part A and Part B: Time to reach maximum observed concentration (tmax) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  tmax of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A (A1 and A2 only): Time of last observed quantifiable concentration (tlast) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose)
  tlast of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Maximum observed serum (peak) drug concentration (Cmax) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  Cmax of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Maximum observed serum (peak) drug concentration divided by the lung-delivered dose (LDD) [Cmax/D] of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  Cmax/D of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Concentration at the end of the dosing interval (Ctrough) [repeat dose only] of AZD8630 | Pre-dose and Post-dose: Part A- (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  Ctrough of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Partial area under the serum concentration-time curve from 0 to time 24 hours post-dose [AUC(0-24)] of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), and Day 1 for MAD and Part B
  AUC(0-24) of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Partial area under the serum concentration-time curve from 0 to time 24 hours post-dose divided by the LDD [AUC(0-24)/D] of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), and Day 1 for MAD and Part B
  AUC(0-24)/D of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A: Area under the serum concentration curve from zero to the last quantifiable concentration (AUClast) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose)
  AUClast of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A: Area under the serum concentration-time curve from time zero to time of last quantifiable drug concentration divided by the LDD (AUClast/D) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose)
  AUClast/D of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Area under serum concentration-time curve from zero to infinity (AUCinf) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), and Day 1 for MAD and Part B
  AUCinf of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Area under the serum concentration-time curve from time zero extrapolated to infinity divided by the LDD (AUCinf /D) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), and Day 1 for MAD and Part B
  AUCinf /D of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Area under serum concentration-time curve in the dosing interval t (AUCt) of AZD8630 | Pre-dose and Post-dose: Part A- (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  AUCt of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Area under serum concentration-time curve in the dosing interval t divided by the LDD (AUCt/D) of AZD8630 | Pre-dose and Post-dose: Part A- (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  AUCt/D of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Terminal rate constant (λz) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  λz of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  t1/2λz of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Mean residence time of the unchanged drug in the systemic circulation (MRTinf) of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  MRTinf of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Apparent total body clearance of drug from serum after extravascular administration (inhalation administration only) [CL/F] of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  CL/F of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Apparent volume of distribution following extravascular administration based on terminal phase (inhalation administration only) [Vz/F] of AZD8630 | Pre-dose and Post-dose: Part A- (SAD) Days 1 to 4 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1 to 14, Day 28, Day 29, and FU Visit/ ET Visit (10-day post-last dose)
  Vz/F of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Accumulation ratio based upon AUCt [Rac(AUC)] of AZD8630 | Pre-dose and Post-dose: Part A- (MAD) Day 14; Part B- Day 28
  Rac(AUC) of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Accumulation ratio based upon Cmax [Rac(Cmax)] of AZD8630 | Pre-dose and Post-dose: Part A- (MAD) Day 14; Part B- Day 28
  Rac(Cmax) of AZD8630 in healthy participants, including participants of Japanese and Chinese ethnicity will assessed.
Part A and Part B: Number of participants with presence of anti-drug antibodies (ADAs) | Pre-dose: Part A- (SAD) Days 1 to 3 and FU Visit/ET Visit (7-day post-dose), (MAD) Days 1 to 17 and FU Visit/ET Visit (10-day post-last dose); Part B- Days 1, 7, 14, and 28, and FU Visit/ ET Visit (10-day post-last dose)
  Immunogenicity of AZD8630 following single and multiple dose administration will be characterized.
Part B: Change from baseline in fractional exhaled nitric oxide (FeNO) levels | From Screening (Up to days 28 before Day 1) until Day 29 (end of the treatment visit)
  The PD effect of AZD8630 on FeNO versus placebo following daily inhaled AZD8630 will be assessed.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (14):
  - Research Site, Tempe, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Glendale, California
  - Research Site, San Jose, California
  - Research Site, Homestead, Florida
  - Research Site, Miami, Florida
  - Research Site, Boise, Idaho
  - Research Site, White Marsh, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Raleigh, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, El Paso, Texas
- Germany (6):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Wiesbaden
- United Kingdom (4):
  - Research Site, Bradford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home